CLINICAL TRIAL: NCT05670899
Title: Retention of CAD Metallic and Poly Ether Ether Ketone (PEEK) Frameworks in Mandibular Kennedy Class I Cases: a Randomized Clinical Trial
Brief Title: Retention of CAD Metallic and Poly Ether Ether Ketone (PEEK) Frameworks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Magdy Ibrahim, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91122
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Retention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD PEEK frame-work (Experimental): Construction of PEEK framework will be done conventionally by lost wax technique using a vacuum press device. The wax pattern will be invested in a mold using special investment. Then it will be heated and melted to produce a mold into which PEEK will be vacuum pressed. The framework will be fitted on the master cast
  Interventions: Procedure: CAD PEEK frame-work
- CAD metallic frame-work (Active Comparator): A metallic framework will be obtained using the conventional lost wax technique and casting. After de-investing, finishing and polishing, the framework will be fitted on the master cast. Intraoral try in of the framework will be done followed by bite registration record. The next step will be teeth setting and try in. Heat cured acrylic resin denture base will be processed, finished and polished conventionally. The finished removable partial denture will then be checked intraorally for any needed modifications and finally delivered.
  Interventions: Procedure: CAD PEEK frame-work

INTERVENTIONS:
Procedure: CAD PEEK frame-work — Construction of PEEK framework will be done conventionally by lost wax technique using a vacuum press device. The wax pattern will be invested in a mold using special investment. Then it will be heated and melted to produce a mold into which PEEK will be vacuum pressed. The framework will be fitted on the master cast

SUMMARY:
comparing retention of CAD CAM metallic and Poly Ether Ether Ketone (PEEK) partial dentures in Kennedy class I casses

DETAILED DESCRIPTION:
partially edentulous patients with Kennedy class I classification will be recruited for the trial and then randomly distributed on two groups; experimental group will receive CAD CAM PEEK partial denture and control group will receive CAD CAM metallic partial denture. then primary impressions will be made and then mouth preparation followed by secondary impression then scanning of the master cast using extra-oral scanner then designing the partial denture using blender for dental then the frame work will be printed.

then frame work will be processed into either PEEK or Metal according to randomization.

retention will be measured at zero and 3 months.

ELIGIBILITY:
Inclusion Criteria:

- Patients with bilateral free end saddles in the mandible (kennedy class I) with last standing abutment premolar.

2- Opposing dentition is fully intact or restored. 3- Sufficient inter-arch space. 4- Angle's class I maxilla-mandibular relationship.

Exclusion Criteria:

1. Periodontal affection of the abutment teeth.
2. Skeletal mal-relation.
3. Unmotivated patients to maintain adequate oral hygiene to follow up.
4. Patients with neuromuscular and Psychiatric disorders.
5. Systematic disease affecting bone and periodontal health.
6. Insufficient inter-arch space.
7. Patients with physical reasons that could affect follow up.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-20 (Estimated); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
retention | 3 months
  Measurements are performed for each RPD at the time of denture insertion, after one month and three months later. Measurements were carried out using digital force gauge which is an advanced type of force meter device, used to measure tension or compression up to 20 Kg

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Manial, Egypt